CLINICAL TRIAL: NCT06981455
Title: LIFE-NETs (Life Following Excision of Neuroendocrine Tumors): a Multi-institutional Prospective Observational Cohort Study of Quality of Life After Surgery for Neuroendocrine Tumors
Brief Title: Life Following Excision of Neuroendocrine Tumors
Acronym: LIFENETS
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Julie Hallet, Associate Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: SHSC-REB-6147
Record Dates: First submitted 2025-04-23; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine (NE) Tumors; Neuroendocrine Tumor GEP Grade 1-3
Keywords: surgery; quality of life; carcinoid; neuroendocrine
MeSH Terms: conditions — Neoplasms; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resected GEP-NETs: Surgery for resection of NETs, including complete resection and cytoreduction resection, as advised by the treating physician. The extent and timing of surgery is determined by the treating physician.

SUMMARY:
Neuroendocrine tumors (NETs), often seen as "chronic cancer" present a survival paradox with relatively prolonged patient survival despite active disease. Treatment strategies emphasize management over cure, integrating tumor control with quality of life (QOL) considerations. Surgery is a cornerstone of NET management but demands a careful balance between its potential benefits and the morbidity risks. Current literature on post-surgical QOL is limited and non-generalizable, underscoring the need for comprehensive, multi-institutional data to inform surgical decisions.

We will study QOL after surgery for NETs in a prospective multi-institutional international cohort study. Specifically, we aim to 1) describe the post-operative QOL of patients with NETs and 2) identify factors associated with QOL measures after surgery for NETs. This project will be led in partnership by the Susan Leslie Clinic for NETs at Sunnybrook Health Sciences Centre in Toronto, Canada, and the IRCCS San Raffaele ENETS Centre of Excellent in Milan, Italy, and enrol adults undergoing surgery for resection of gastro-entero-pancreatic NETs across 12 North-American and European high-volume NETs surgery centres over a 18-month period. Measures of QOL using the SF-12 Survey, the EORTC-QLQ C30 and GEPNET21 tool, and clinical symptoms assessment, will be captured prior to surgery and at 6, 12, 24, and 36 months after surgery. Mixed linear regression models with random intercepts to account for longitudinal data correlation and individual variability will be used to analyze the QOL measures over time. Patient and service users engagement (PSUE) will be integrated throughout the study continuum.

This project will fill the knowledge gap in QOL after surgery for NETs, with a view to support better-informed surgical decisions and patient-centred care. The prospective, multi-institutional, and international design promises a comprehensive understanding of the impact of surgery on patient's lives, potentially shaping management pathways globally.

DETAILED DESCRIPTION:
Background

Neuroendocrine neoplasms (NENs) are a unique group of malignancies distinguished by their more indolent biology and endocrine secretion.1 Because of indolent biology, patients with well-differentiated NENs (neuroendocrine tumors - NETs) can experience prolonged survival even in the presence of active disease, with up to 50% at 10 years, and may be considered a "chronic cancer". Unlike other malignancies, the goals of therapy for NETs are largely focused on control over cure. Rather than focusing solely on tumor eradication, treatment aims for long-term management that encompasses both tumor and endocrine control as well as prevention of loco-regional complications from tumor deposits.

Surgery holds a pivotal role in the management of NETs, both for loco-regional and advanced disease with distant metastases.4 As an initial intervention, surgery serves a dual purpose. First, it acts as a primary treatment modality for achieving tumor and endocrine control. Second, by reducing the tumor burden surgically, it can have therapy-sparing effects whereby it can delay the need for subsequent lines of therapy, which often come with their own side effects and complications. This is especially important in the treatment of a chronic cancer where patients are expected to require ongoing management in the long-term.

However, the decision to opt for surgery is not straightforward. There's an intricate balance that is needed between the potential benefits of surgery and the potential risks of post-surgical morbidity. Indeed, some have voiced concerns that the potential risks and costs associated with surgical morbidity may outweigh the benefits.

A considerable gap in our understanding of the benefits of surgery for NETs is the lack of data regarding patients' quality of life post-surgery. The majority of existing research on this topic either adopts a retrospective approach or lacks the application of standardized, validated tools for assessment. Recently, a single-centre study analyzed a cohort of 31 patients undergoing surgical treatment for small bowel and pancreatic NETs, including 46% of patients with metastases. Using the SF-12 questionnaire, that study reported improvements in both mental and physical health at 12 months post-surgery compared to pre-operative levels. The largest improvements were observed in patients with larger primary tumors, metastatic disease, or those who received systemic therapy after surgery. However, the study's limited sample size and single-centre design significantly restrict its generalizability.

To better position the role of surgery in the management of NETs, it is imperative that we bridge this knowledge gap with robust, multi-institutional prospective studies. This proposal seeks to address this need, ensuring that surgical decisions are made with a comprehensive understanding of patients' quality of life following surgery.

Objectives

In a prospective multi-institutional international cohort of patients, we aim to

1. Describe quality of life (QOL)measures following surgery for NETs;
2. Identify factors associated with QOL measures following surgery for NETs.

Sampling and recruitment

A convenience sample of patients will be recruited from surgery clinics at participating centres. Recruitment will take place over 18 months and follow-up continued for 36 months for all patients.

Analysis

We will summarize sociodemographic and clinical characteristics as well as outcomes values using descriptive statistics with means and standard deviation (SD) or median and inter-quartile range (IQR) for continuous variables, and absolute number (n) with percentage (%) for categorical variables. Boxplots and histograms will be used to present the distribution of outcomes values at each timepoint.

We will analyze the longitudinal outcomes values (score) using mixed linear regression models with random intercept for patients to model the trajectory of scores after surgery. The models will estimate the relative change in a patient's scores over time while adjusting for potential confounders. This approach accounts for the fact the observations are not independent since the repeated measures come from the same patients over time. This model will allow to account for random effects as individuals will be sampled at random from a population and may exhibit random variation between themselves. Such variability is expected and likely to represent natural heterogeneity among individuals because of factors difficult to measure, such as prior experiences or personality traits. The model will also address correlation within repeated measures from the same individual over time. We hypothesize that the change in scores over time will be non-linear; therefore, we will examine this relationship and plan to include a quadratic term for time to better model the non-linear relationship if appropriate. Using those models, we will plot the expected trajectory of patients over time with 95% confidence bands.

We have planned to explore differences in outcomes scores trajectories based on key sociodemographic and clinical factors by including interaction terms between time and key factors of interest defined a priori. These factors are: age (<70 years old vs >70 years old), sex (male vs. female), primary tumor site (pancreas vs. midgut), grade (grade 1 vs. grade 2), and type of surgery (pancreatectomy, small bowel resection, liver resection).

All analyses will be two-sided, with statistical significance set at p<0.05.

Interim analysis

An a priori interim analysis will be conducted 12 months after the end of the enrollment period, to analyze QOL data at 12 months after surgery. The final analysis will be conducted 36 months after the end of the recruitment period.

Patient and service users' engagement

Patient and service users' engagement (PSUE) is known to enhance the relevance, validity, quality, and applicability of research. We have planned for integrated engagement throughout the study continuum using the PSUE framework. Consistent with The Change Foundation decision tool, thank you notes and gift certificates will be sent to all participants engaged in the study. We will assess the quality of our PSUE using the Public and Patient Engagement Evaluation Tool (PPEET). PSUE participants will be recruited via patient advocacy associations upon initiation of the project.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Diagnosis of well-differentiated grade 1 to 3 NETs via histopathology (biopsy) or imaging (measurable tumor on CT or MRI with avidity on SSTR-PET scan).
* Consents to surgery for resection of localized, loco-regional, or metastatic gastro-enteric (midgut) and pancreatic neuroendocrine tumor (GEP-NET).

Exclusion Criteria:

* Pre-operative diagnosis of neuroendocrine carcinoma on histopathology (biopsy) or imaging (measurable tumor on CT or MRI with avidity on FDG-PET scan and no avidity on SSTR-PET scan).
* Declines surgery.
* Unable to respond to study questionnaires (not proficient in local language).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for resection of gastro-entero-pancreatic neuroendocrine tumors.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Within 30 days before surgery (pre-operative) and at 6, 12, 24 and 36 months after surgery
  Quality of life will be measured by the 12-item short-form quality of life survey (SF-12).
  The SF-12 is a validated tool that evaluates limitations in physical, social, and work activities due to physical or emotional problems to provide a measure of functional health and wellbeing. It evaluates 8 domains of quality of life: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. This survey has been tested both in the general population and in a variety of diseases, and is able to reflect changes in quality of life over time. Two composite scores are obtained from answers to the SF-12: the physical composite score (PCS) and the mental composite score (MCS). Average PCS and MCS for the general population are 50 points each with a standard deviation of 10 points. The SF-12 score goes from 0 to 100, with higher scores indicating better performance.

OTHER OUTCOMES:
Self-reported patient symptoms | 6, 12, 24 and 36 months after surgery
  Patients' description of their symptoms will also be recorded at the pre-operative visit and re-examined and tracked at each follow-up assessment as improved, unchanged, or worsened as per patients' assessment.
QoL questionnaire EORTC-QLQ C30 | within 30 days of surgery and at 6, 12, 24 and 36 months after surgery
  The EORTC-QLQ C30 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire) is a validated tool for use in patients with cancer and is widely used and accepted in cancer research. The GEPNET21 is a supplement to the QLQ-C30 which asks specific NET questions and has been validated in patients with NETs. It is recommended that both be used together.
  Using a linear transformation to standardise the raw score, the scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No